CLINICAL TRIAL: NCT02629094
Title: Cardiometabolic Effects of Eplerenone in HIV Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160030; 16-I-0030
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2017-09

CONDITIONS: Cardiac Steatosis; Hepatic Steatosis
Keywords: Hepatic Steatosis; Cardiac Steatosis; Aldosterone; Eplerenone; Mineralcorticoid Receptor
MeSH Terms: conditions — Fatty Liver | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Intervention: Eplerenone will be administered for 6 months as follows: 25 mg once daily for 1 week and then 50 mg once daily for the remainder of the study.
  Interventions: Drug: Inspra /Eplerenone

INTERVENTIONS:
Drug: Inspra /Eplerenone — Eplerenone is provided as 25- or 50-mg tablets that are to be taken orally. Subjects will be dosed at 25 mg daily for 1 week, and then 50 mg daily for 23 weeks. The total duration of dosing for each subject is 24 weeks.

SUMMARY:
Background:

People with human immunodeficiency virus (HIV) are at a high risk of getting visceral or deep belly fat. Visceral fat can cause health problems like heart or liver disease. Researchers want to see if a blood pressure drug can help by blocking a hormone in the body.

Objective:

To see if eplerenone reduces fat stored in the heart muscle and liver in people with HIV and increased visceral fat.

Eligibility:

Adults ages 18 75 with HIV and increased waist circumference. Increased waist circumference is defined as more than 40 inches in men and more than 35 inches in women.

Design:

Participants will be screened with:

Physical exam

Medical history

Blood tests

Measurements of hips, waist, legs, arms, shoulders, and neck

Magnetic resonance imaging (MRI) scan. They will lie on a table that slides into a machine.

Electrocardiogram (EKG) to measure heart electrical activity

Transient elastography, a special ultrasound to measure liver tissue stiffness

A small piece their liver collected (optional)

Participants will have a baseline visit:

Physical exam

Medical history

Blood tests

DEXA scan to measure body fat, muscle mass, and bone density. Participants will lie on a table while a very small dose of x-rays goes through the body.

Resting energy expenditure (REE). This measures the amount of oxygen breathed in and carbon dioxide breathed out.

Participants will get a 1-week supply of eplerenone. They will take one pill per day.

Participants will have a follow-up visit 1 week later. They will have:

Physical exam

Medical history

Blood tests

23-week supply of eplerenone

Participants will have 5 more follow-up visits.

Participants will have a final study visit, repeating many of the screening and baseline tests.

DETAILED DESCRIPTION:
HIV-infected individuals are at higher risk than uninfected people for developing cardiovascular disease. Visceral adipose tissue is also increased in HIV-infected people compared to uninfected individuals. Animal studies suggest that blockade of the mineralocorticoid receptor (MR) may have beneficial effects on cardiovascular and metabolic parameters via inhibition of adipocyte differentiation and triglyceride accumulation. We will examine the effects of the MR antagonist eplerenone (50 mg daily) on HIV-infected adults with abdominal fat accumulation in a 24-week, open-label, proof-of-concept study. Magnetic resonance imaging will be conducted at screening and the final study visit to evaluate cardiac and hepatic steatosis. We anticipate that blocking the effects of increased aldosterone secretion with eplerenone will significantly reduce intramyocardial lipid content and hepatic steatosis in this population. These effects may be accompanied by decreases in visceral adipose tissue, and improvements in dyslipidemia and inflammation, thereby improving cardiovascular health.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Increased waist circumference on the basis of National Cholesterol Education Program guidelines (> 102 cm in men and > 88 cm in women)
  2. Hepatic steatosis established by hepatic MRI greater than or equal to 5% and/or liver biopsy within the last 12 months
  3. HIV-infected, HIV viral load < 50 copies/mL and no change in ART regimen for at least 3 months
  4. Age greater than or equal to 18 and less than or equal to 75 years
  5. Agree to have samples stored for future research

EXCLUSION CRITERIA:

1. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m^2, serum creatinine > 1.5 mg/dL
2. Serum potassium > 5.5 mEq/L, alanine aminotransferase > 2.5 times the upper limit of normal, hemoglobin (Hgb) < 11 g/dL
3. Uncontrolled hypertension: systolic blood pressure greater than or equal to 160 mm Hg or diastolic blood pressure greater than or equal to 100 mm Hg
4. A blood pressure < 90mmHg systolic or < 50mm Hg diastolic
5. Screening EKG with a significant heart block (e.g. PR > 300 ms) or an EKG determined significant by Cardiology consult.
6. Current hepatitis C infection, unless there has been a sustained virologic response for at least 12 months
7. Type 2 diabetes with microalbuminuria
8. Current or prior steroid use within past 6 months (except short-course or single-dose administration). Stable use of inhaled or nasal steroids are allowed.
9. Use of angiotensin converting enzyme (ACE) inhibitors, angiotensin reporter blockers (ARBs), potassium-sparing diuretics, and other medications that may increase the risk of hyperkalemia
10. Use of potassium supplementation or other medications known to increase potassium
11. Concomitant use of strong inhibitors and/or inducers ofof cytochrome P450 isozyme (CYP)3A4
12. If receiving testerone, estrogen or progesterone therapy, must be on a stable dose for at least 3 months.
13. Current use of growth hormone or growth hormone-releasing hormone
14. Current serious viral, bacterial, or other infection (excluding HIV)
15. Current active substance abuse/dependence
16. Substantial history of cardiovascular disease, including prior myocardial infarction (MI), congestive heart failure, or stroke
17. Contraindication to MRI
18. Pregnant or planning to become pregnant
19. Breastfeeding
20. Any condition that, in the opinion of the PI, may substantially increase the risk of participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12-02; Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Hadigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Triant VA, Lee H, Hadigan C, Grinspoon SK. Increased acute myocardial infarction rates and cardiovascular risk factors among patients with human immunodeficiency virus disease. J Clin Endocrinol Metab. 2007 Jul;92(7):2506-12. doi: 10.1210/jc.2006-2190. Epub 2007 Apr 24. PMID 17456578
- [Background] Hirata A, Maeda N, Hiuge A, Hibuse T, Fujita K, Okada T, Kihara S, Funahashi T, Shimomura I. Blockade of mineralocorticoid receptor reverses adipocyte dysfunction and insulin resistance in obese mice. Cardiovasc Res. 2009 Oct 1;84(1):164-72. doi: 10.1093/cvr/cvp191. Epub 2009 Jun 8. PMID 19505930
- [Background] Suzuki J, Iwai M, Mogi M, Oshita A, Yoshii T, Higaki J, Horiuchi M. Eplerenone with valsartan effectively reduces atherosclerotic lesion by attenuation of oxidative stress and inflammation. Arterioscler Thromb Vasc Biol. 2006 Apr;26(4):917-21. doi: 10.1161/01.ATV.0000204635.75748.0f. Epub 2006 Jan 19. PMID 16424347
- [Result] Chaudhury CS, Purdy JB, Liu CY, Morse CG, Stanley TL, Kleiner D, Hadigan C. Unanticipated increases in hepatic steatosis among human immunodeficiency virus patients receiving mineralocorticoid receptor antagonist eplerenone for non-alcoholic fatty liver disease. Liver Int. 2018 May;38(5):797-802. doi: 10.1111/liv.13734. Epub 2018 Mar 31. PMID 29509992

RESULTS

PARTICIPANT FLOW:
Groups:
- Eplerenone: Eplerenone 25mg once/day for one week; 50mg once/day 23 weeks
Period: Overall Study
Arm/Group | Eplerenone
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All screened participants were evaluated for baseline data, of which 5 were eligible to start.
Arm/Group | Eplerenone
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Cardiac Steatosis: Mean Change in Intraventricular Septum Percentage of Lipid by MR Spectroscopy.
Description: Mean change in intraventricular septum percentage of lipid by MR spectroscopy. This was calculated by subtracting the baseline intraventicular septum percentage value of lipid from the week 24 intraventicular septum percentage value of lipid by MR spectroscopy.
Time Frame: 24 weeks
Population: Analyses included participants who completed 24 weeks on study drug eplerenone.
Measure: Mean (Standard Deviation); unit: percentage of lipid
Arm/Group | Eplerenone
Number analyzed (Participants) | 5
percentage of lipid | -0.33 (4.3)

2. Primary Outcome: Improvement of Hepatic Steatosis: Mean Change in Hepatic Percentage of Lipid by MR Spectroscopy
Description: Mean change in hepatic percentage of lipid by MR spectroscopy. This was calculated by subtracting the baseline hepatic percentage value of lipid from the week 24 hepatic percentage value of lipid by MR spectroscopy.
Time Frame: 24 weeks
Population: Analyses included participants who completed 24 weeks on study drug eplerenone.
Measure: Mean (Standard Deviation); unit: percentage of lipid
Arm/Group | Eplerenone
Number analyzed (Participants) | 5
percentage of lipid | 13 (7.3)

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Eplerenone
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eplerenone (N=5)
Acute sinusitis (Infections and infestations) | 1 (1)
Blood bicarbonate decreased (Investigations) | 2 (2)
Blood calcium increased (Investigations) | 1 (3)
Blood creatinine increased (Investigations) | 1 (2)
Blood glucose increased (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 2 (2)
Blood potassium decreased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT02629094/Prot_SAP_000.pdf